CLINICAL TRIAL: NCT01546532
Title: A Multicenter, Randomized, Double-blind, Parallel Group, Placebo-controlled Study to Evaluate the Renal Hemodynamic Effects of RLX030 and Placebo Infused for 24 Hours in Subjects With Chronic Heart Failure (CHF)
Brief Title: Renal Hemodynamic Effects of RLX030A in Subjects With Chronic Heart Failure (CHF)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CRLX030A2202; 2011-001588-37 (EudraCT Number)
Record Dates: First submitted 2012-03-02; First posted 2012-03-07 (Estimated); Last update posted 2020-12-19 (Actual); Status verified 2013-02

CONDITIONS: Chronic Heart Failure (CHF)
Keywords: Heart failure; RLX030; hemodynamics; cardiovascular diseases
MeSH Terms: conditions — Heart Failure; Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- RLX030 (Experimental): RLX030 as intravenous infusion for 24 hours.
  Interventions: Drug: RLX030
- Placebo (Placebo Comparator): Placebo as intravenous infusion for 24 hours.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: RLX030 — RLX030 as intravenous infusion for 24 hours.
  Arms: RLX030
Drug: Placebo — Intravenous infusion of Placebo over 24 hours
  Arms: Placebo

SUMMARY:
This study will assess the renal hemodynamic effect of RLX030 infusion in subjects with chronic heart failure. In addition safety and effects on renal function and biomarkers will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent must be obtained before any assessment is performed.
* Male and female heart failure patients with body weight <160 kg, on standard therapy including a stable dose of furosemide 40-240 mg/day orally (p.o). or equivalent dose of loop diuretics, reduced systolic function (LVEF ≤ 45% measured within the past 6 months), BNP ≥ 100 pg/mL or NT-pro-BNP of ≥ 400 pg/mLNYHA Class II or III, and worsening symptoms, e.g. fatigue, dyspnea, breathlessness within 3 months
* Mild to moderate renal impairment

Exclusion criteria:

* Systolic blood pressure (SBP) < 110 mm Hg at the time of randomization
* Administration of intravenous radiographic contrast agent within 72 hours prior to randomization or acute contrast-induced nephropathy at the time of randomization
* Current use of non-steroidal antiinflammatory drugs (NSAIDs)
* Current or planned (through the completion of study drug infusion) treatment with any i.v. therapies, including vasodilators (including nesiritide), positive inotropic agents, vasopressors, levosimendan, or mechanical support (intra-aortic balloon pump, endotracheal intubation, mechanical ventilation, or any ventricular assist device).
* Clinically significant hepatic impairment defined as hepatic encephalopathy of any degree or total bilirubin > 50 μmol/l (3 mg/dl) or, if patient is not on warfarin therapy, INR > 2.0 (or Prothrombin Time > 2 * ULN)

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2012-02; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in renal plasma flow (RPF) measured by Para-aminohippuric acid (PAH) clearance in subjects with CHF after 24 hours intravenous (i.v) infusion of RLX030 | Baseline, during and after the end of 24 hours infusion
  Serial blood and urine collections over time for determination of PAH and its clearance respectively
Change from baseline in glomerular filtration rate (GFR) as measured by Iothalamate (IOTH) clearance in subjects with CHF after 24 hours i.v. infusion of RLX030 | Baseline, during and after the end of 24 hours infusion
  Serial blood and urine collections over time for determination of IOTH and its clearance respectively

SECONDARY OUTCOMES:
Change from baseline in filtration fraction (FF) in subjects with CHF after 24 hours infusion of RLX030 | Baseline, during and after the end of 24 hours of infusion
  The filtration fraction (FF) is derived as the ratio of GFR divided by RBF in percent.
Change over time in Diuresis | During 24 hours of infusion and after the end of the infusion
  Urine samples will be collected for analyses.
Change over time in calculated creatinine clearance | During 24 hours of infusion and after the end of the infusion
  Urine samples will be collected for analyses.
Change over time on fractional sodium excretion(natriuresis) | During 24 hours of infusion and after the end of the infusion
  Urine samples will be collected for analyses.
Central aortic systolic pressure-time curve | During 24 hours of infusion and after the end of the infusion
  A cuff will be used for a brachial blood pressure measurement and a wrist sensor for arterial pulse waveforms
Radial augmentation index-time curve | During 24 hours of infusion and after the end of the infusion
  A cuff will be used for a brachial blood pressure measurement and a wrist sensor for arterial pulse waveforms
Number of patients with adverse events, serious adverse events and death | During 24 hours of infusion and after the end of the infusion
  Monitoring of adverse events, serious adverse events and death from screening to end of study
Pharmacokinetics of RLX030: area under the serum concentration-time curve from time zero to infinity (AUCinf)Time | During 24 hours of infusion and for 24 hours after the end of infusion
  Blood will be collected from an indwelling catheter.
Pharmacokinetics of RLX030: area under the serum concentration-time curve from time zero to the time of the last quantifiable concentration (AUClast) | During 24 hours of infusion and for 24 hours after the end of infusion
  Blood will be collected from an indwelling catheter.
Pharmacokinetics of RLX030: serum concentration over 20 hours of infusion (C24h) | During 24 hours of infusion and for 24 hours after the end of infusion
  Blood will be collected from an indwelling catheter.
Pharmacokinetics of RLX030: terminal elimination half-life (T1/2)following intravenous administration | During 24 hours of infusion and for 24 hours after the end of infusion
  Blood will be collected from an indwelling catheter.
Pharmacokinetics of RLX030: mean residence time (MRT)intravenous administration | During 24 hours of infusion and for 24 hours after the end of infusion
  Blood will be collected from an indwelling catheter.
Pharmacokinetics of RLX030: volume of distribution at steady state (Vss) following intravenous administration | During 24 hours of infusion and for 24 hours after the end of infusion
  Blood will be collected from an indwelling catheter.
Pharmacokinetics of RLX030: systemic clearance from serum (CL) following intravenous administration(natriuresis) | During 24 hours of infusion and for 24 hours after the end of infusion
  Blood will be collected from an indwelling catheter.
Corrected QT (QTc) Interval Using Fridericia's and Bazett's Formula | Baseline, during the 24 hours of infusion and after the end of the infusion
  Continuous 12 lead Holter ECG monitoring for extraction of ECGs and analysis

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (14):
- Novartis Investigative Site, Baltimore, Maryland, United States
- Germany (4):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Erlangen
  - Novartis Investigative Site, Göttingen
  - Novartis Investigative Site, Hamburg
- Netherlands (3):
  - Novartis Investigative Site, Deventer
  - Novartis Investigative Site, Groningen
  - Novartis Investigative Site, Sneek
- Poland (6):
  - Novartis Investigative Site, Grodzisk Mazowiecki
  - Novartis Investigative Site, Katowice
  - Novartis Investigative Site, Krakow
  - Novartis Investigative Site, Lublin
  - Novartis Investigative Site, Warsaw
  - Novartis Investigative Site, Wałbrzych

REFERENCES:
- [Derived] Voors AA, Dahlke M, Meyer S, Stepinska J, Gottlieb SS, Jones A, Zhang Y, Laurent D, Slart RH, Navis GJ. Renal hemodynamic effects of serelaxin in patients with chronic heart failure: a randomized, placebo-controlled study. Circ Heart Fail. 2014 Nov;7(6):994-1002. doi: 10.1161/CIRCHEARTFAILURE.114.001536. Epub 2014 Oct 6. PMID 25286914
- See also: Results for CRLX030A2202 from the Novartis Clinical Trials website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=10684